CLINICAL TRIAL: NCT05858229
Title: A Phase 1B Study of Intralesional Injection of RP1 in Patients With Resectable Cutaneous SCC
Brief Title: Neo-adjuvant Treatment for Squamous Cell Carcinoma Using Direct Tumor Injection With RP1.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sherrif Ibrahim (Other)
Responsible Party: Sponsor-Investigator, Sherrif Ibrahim, Principal Investigator, Rochester Dermatologic Surgery
Organization: Rochester Dermatologic Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST2021-RP1-08
Record Dates: First submitted 2023-04-17; First posted 2023-05-15 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma; RP1
Keywords: squamous cell carcinoma; RP1; intralesional treatment; non-surgical option
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients will receive RP1 via direct intratumoral (IT) injection into superficial cutaneous solid tumors to assess the safety and tolerability as well efficacy of RP1 treatment. The primary efficacy population is up to 12 evaluable patients with resectable CSCC.
  Interventions: Drug: RP1

INTERVENTIONS:
Drug: RP1 — Recombinant Herpes Simplex Virus Type 1 - hGM CSF/GALV-GP-R-

SUMMARY:
This is a Phase 1b, single-center, open-label study, evaluating efficacy and safety of RP1 for the treatment of resectable cutaneous Squamous Cell Carcinoma in up to 12 evaluable patients. In this study, patients will receive RP1 via direct intratumoral (IT) injection into superficial cutaneous solid tumors to assess the safety and tolerability as well efficacy of RP1 treatment. The primary efficacy population is up to 12 evaluable patients with resectable CSCC. The enrollment of patients with CSCC will determine study duration.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent prior to any study procedures and the willingness and ability to comply with all aspects of the protocol.
* Male or female ≥ 18 years of age on the day of signed informed consent.
* Patients must be treatment naïve in the target lesion(s).
* Patients for whom surgical treatment of lesions is clinically indicated.
* At least one measurable histologically confirmed cutaneous tumor of ≥ 1.0 cm in longest diameter and ≤ 3.0 cm with clinically visible residual tumor. More than one tumor may be treated including newly diagnosed lesions.
* ECOG performance status ≤ 1.
* Adequate hepatic function, including both of the following:
* Adequate hematologic function
* Adequate coagulation parameters, including both of the following:
* Anticipated life expectancy > 2 years
* Have provided either formalin-fixed, paraffin-embedded (FFPE) tissue block or unstained tumor tissue sections, obtained within four months prior to enrollment, with an associated pathology report,. Biopsy can be either by punch or shave method.. A fresh biopsy is required at screening if an archival biopsy (within four months prior to enrollment) is not available.

Exclusion Criteria:

* Prior treatment with an oncolytic therapy or intratumoral immunotherapy (e.g. TLR agonists, etc.).
* Patients with known visceral metastases.
* Active significant herpetic infections or prior complications of HSV-1 infection (e.g., herpetic keratitis or encephalitis). Patients who require intermittent or chronic use of systemic (oral or IV) antiviral agents with known antiherpetic activity (e.g., acyclovir, valacyclovir, famciclovir, ganciclovir, valganciclovir). Note: Patients with sporadic cold sores may be enrolled as long as no active cold sores are present at the time of first dose of RP1.
* Had systemic infection requiring IV antibiotics or other serious infection within 14 days prior to dosing.
* Patients with an active, known, or suspected autoimmune disease that requires systemic immunosuppressive treatment. Patients with vitiligo, childhood asthma that has resolved, type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, or psoriasis that does not require systemic treatment are permitted to enroll.
* Patients with a history of any positive test result for hepatitis B virus (HBV) or hepatitis C virus (HCV) indicating the presence of the virus, e.g., hepatitis B surface antigen [HBsAg] positive or hepatitis C antibody (anti-HCV) positive (except if HCV RNA negative), or human immunodeficiency virus (HIV) positive. Patients with a history of HBV or HCV infection must have undetectable viral load within three months of study entry. (Note: No testing for HBV, HCV, or HIV is required unless mandated by local health authorities).
* Had clinically significant cardiovascular disease within 6 months from first dose of study drug, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction or stroke/transient ischemic attack or significant cardiac arrhythmias associated with hemodynamic instability.
* Radiation therapy within 14 days of first dose of RP1, or topical therapy within 30 days of RP1, is not allowed. The patient must have recovered from all AEs due to previous therapies to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 5.0) Grade 1 or baseline. Participants with unresolved radiation-induced xerostomia are eligible.
* Documented history of allergic reactions or acute hypersensitivity reaction attributed to RP1 or to any of the excipients.
* Patients with solid organ transplantation
* Tumors for which margins are not well defined, either clinically or based on pathologic report (Ill-defined tumors).
* Tumors where invasion beyond the subcutaneous fat is suspected
* Any co-morbidity, physical examination finding, metabolic dysfunction, or clinical laboratory abnormality that, in the opinion of the investigator, renders the patient unsuitable for participation due to safety risks and/or potential to affect interpretation of results of the study.
* Treatment with botanical preparations (e.g., herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within two weeks prior to the first dose of RP1 and throughout the study as per Section 5.10.2.
* Any active malignancy within three years of the date of first planned dose of RP1, except for the specific cancer under investigation in this study and tumors with negligible risk of metastasis or death, squamous cell carcinoma in situ (SCCIS), basal cell carcinoma (BCC) or other small CSSS, melanoma in situ, carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, low-risk early stage prostate adenocarcinoma (T1T2aN0M0), Gleason score ≤ 6, and prostate specific antigen (PSA) ≤ 10 ng/mL) for which the management plan is active surveillance, or prostate adenocarcinoma with biochemical-only recurrence with documented PSA doubling time of > 12 months for which the management plan is active surveillance. Patients with hematologic malignancies are excluded, except for patients with chronic lymphocytic leukemia (CLL) who are considered stable and not on active treatment.
* Any acute or chronic psychiatric problems, alcohol abuse, or substance abuse disorders that, in the opinion of the investigator, would interfere with the patient's ability to comply with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate degree of pathologic response at 16 weeks. | 16 weeks
  The proportion of patients with pathologic complete response (pCR) per Immune-Related Pathologic Response Criteria' (irPRC) criteria: 0% residual viable tumor (RVT)] remaining in post-therapy specimen (no signs of cancer) in tissue samples removed during surgery.

SECONDARY OUTCOMES:
Evaluate the duration of response | 2 years
  To estimate duration of response (DOR) for CSCC and all patients treated, by investigator review.
Evaluate presence of disease | 2 years
  To estimate the progression-free (PFS) for CSCC and all patients treated.
To estimate the complete response (CR) rate | 2 years
  Estimate the complete response (CR) rate for CSCC and all patients treated.
To evaluate the disease control rate (DCR) | 2 years
  To evaluate the disease control rate (DCR) for CSCC and all patients treated.

OTHER OUTCOMES:
Survival rate evaluation | 1 year
  To evaluate efficacy by one-year disease free survival (DFS) rates in CSCC and all patients treated, according to investigator review

CONTACTS AND LOCATIONS:
Overall Officials: Catherine VanHooft, HT, Study Director — Rochester Dermatologic Surgery
Locations (1):
- Rochester Dermatologic Surgery, Victor, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bateman A, Bullough F, Murphy S, Emiliusen L, Lavillette D, Cosset FL, Cattaneo R, Russell SJ, Vile RG. Fusogenic membrane glycoproteins as a novel class of genes for the local and immune-mediated control of tumor growth. Cancer Res. 2000 Mar 15;60(6):1492-7. PMID 10749110
- [Background] Bateman AR, Harrington KJ, Kottke T, Ahmed A, Melcher AA, Gough MJ, Linardakis E, Riddle D, Dietz A, Lohse CM, Strome S, Peterson T, Simari R, Vile RG. Viral fusogenic membrane glycoproteins kill solid tumor cells by nonapoptotic mechanisms that promote cross presentation of tumor antigens by dendritic cells. Cancer Res. 2002 Nov 15;62(22):6566-78. PMID 12438252
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Patel IJ, Rahim S, Davidson JC, Hanks SE, Tam AL, Walker TG, Wilkins LR, Sarode R, Weinberg I. Society of Interventional Radiology Consensus Guidelines for the Periprocedural Management of Thrombotic and Bleeding Risk in Patients Undergoing Percutaneous Image-Guided Interventions-Part II: Recommendations: Endorsed by the Canadian Association for Interventional Radiology and the Cardiovascular and Interventional Radiological Society of Europe. J Vasc Interv Radiol. 2019 Aug;30(8):1168-1184.e1. doi: 10.1016/j.jvir.2019.04.017. Epub 2019 Jun 20. No abstract available. PMID 31229333
- [Background] Simpson GR, Han Z, Liu B, Wang Y, Campbell G, Coffin RS. Combination of a fusogenic glycoprotein, prodrug activation, and oncolytic herpes simplex virus for enhanced local tumor control. Cancer Res. 2006 May 1;66(9):4835-42. doi: 10.1158/0008-5472.CAN-05-4352. PMID 16651439